CLINICAL TRIAL: NCT03602885
Title: EL CENTRO: Engaging Latinos in the Center of Cancer Treatment Options - RCT of Usual Chemotherapy Educational Tools Versus Investigational Chemotherapy Educational Tools
Brief Title: EL CENTRO: Engaging Latinos in the Center of Cancer Treatment Options
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrea Enzinger, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-128; U54CA156732-06A1 (NIH)
Record Dates: First submitted 2018-07-09; First posted 2018-07-27 (Actual); Results first posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Metastatic Pancreatic Cancer; Unresectable Pancreatic Cancer; Metastatic Colorectal Cancer
Keywords: Gastrointestinal Cancer; cancer; palliative; chemotherapy; metastatic; colorectal; pancreatic; communication; informed consent; video; education; oncology; patient-centered; outcomes research
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms; Gastrointestinal Neoplasms; Neoplasms; Neoplasm Metastasis; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy education intervention arm (Experimental): Patients randomized to the chemotherapy education intervention (CEI) arm will be given regimen specific written and video chemotherapy educational materials developed by the study team. The treating oncologist will identify which chemotherapy regimen(s) are being considered, in order to select the appropriate chemotherapy educational tool(s) to give the patient. The patient may be given more than one CEI tool if they are considering more than one regimen. Patients randomized to the intervention arm may receive the intervention in addition to OR in place of the standard institutionally approved chemotherapy information sheets (both are acceptable); this is at the discretion of the treating site or the treating physician.
  Interventions: Behavioral: Chemotherapy education intervention (CEI)
- Usual chemotherapy education arm (Active Comparator): Patients randomized to the usual chemotherapy education (CE) arm will undergo the standard institutional practice of chemotherapy education. The oncologist may also choose to give the patient the institutionally approved chemotherapy information sheets according to site-specific policies and clinical practice.
  Interventions: Behavioral: Usual chemotherapy education (CE)

INTERVENTIONS:
Behavioral: Usual chemotherapy education (CE) — Standard chemo education will given per hospital guideline
  Arms: Usual chemotherapy education arm
Behavioral: Chemotherapy education intervention (CEI) — Video, booklet, and website educational materials
  Arms: Chemotherapy education intervention arm

SUMMARY:
The objective of this study is to improve the chemotherapy decision making process for Latinos with advanced gastrointestinal cancers. In this study Latinos who are considering 1st line chemotherapy for newly diagnosed advanced colorectal or pancreatic cancer will be randomized to usual care or to usual care supplemented by a Spanish/English language multimedia chemotherapy educational intervention. Primary informal caregivers will also be invited to participate.

This research study is evaluating if a new set of educational materials will improve the treatment decision-making process for Latinos with advanced gastrointestinal cancers. This research study will involve about 154 patients and 154 caregivers.

DETAILED DESCRIPTION:
There is growing evidence of racial/ethnic disparities in the quality of communication between oncologists and Latinos with cancer. These communication disparities are evidenced by gaps in Latino's understanding of their condition and treatment options, and by worse satisfaction with provider communication. Limited English proficiency and health literacy are very common among Latinos, yet few interventions have been developed to help Latino cancer patients better understand their condition and treatment options.

In this study the investigators have partnered with Latino patients, providers, and researchers to develop a Spanish/English language intervention aimed at better informing Latinos with advanced gastrointestinal cancers about the risks and benefits of their chemotherapy options. Specifically, the intervention consists of a dual language, regimen-specific suite of videos and booklets explaining the most common chemotherapy options used to treat advanced colorectal cancer and advanced pancreatic cancer. The videos feature Latino patients describing their experiences on treatment, as well as clinicians describing factual information about treatment risks, benefits, and alternatives.

In this study, self-identifying Hispanic/Latino patients with metastatic colorectal cancer, locally advanced and metastatic pancreatic cancer considering treatment with first line chemotherapy will be randomized to the usual care, or to usual care supplemented by access to the relevant chemotherapy educational materials. Caregivers will also be enrolled on the study. Participants will be surveyed at baseline, 2-weeks post-treatment initiation, 2-3 months post-treatment initiation, and 4-6 months post-treatment initiation regarding their understanding of chemotherapy risks and benefits, decisional conflict, and other metrics of informed decision-making.

ELIGIBILITY:
Patient Inclusion Criteria:

* Self-identify as Hispanic/Latino
* Has been diagnosed with metastatic colorectal cancer (mCRC) OR locally advanced pancreatic cancer (LAPC) OR metastatic pancreatic cancer (mPC) AND is making a decision regarding treatment with 1st line palliative chemotherapy
* Treating oncologist has recommended consideration of one or more of the regimens for which we have developed chemotherapy educational (CEI) toolkits

  * For mCRC: FOLFOX, FOLFOX + bevacizumab, FOLFIRI, FOLFIRI + bevacizumab
  * For LAPC or mPC: FOLFIRINOX, Gemcitabine, or Gemcitabine + nab-paclitaxel
  * Patients who are also considering treatment on a clinical trial of one of these regimens +/- an investigational agent would still be eligible, so long as the treating MD believes to the content of the CEI to be relevant to the trial regimen.
* Planning to receive treatment at the enrolling site
* Age ≥ 21
* English or Spanish proficient

Caregiver Inclusion Criteria:

* Caregivers of eligible patient participants
* Age ≥ 21
* English or Spanish proficient

Exclusion Criteria:

* For mCRC patients: Patients with oligometastatic disease who have a definitive plan for curative surgical resection are not eligible.
* Significant delirium/dementia as judged by the treating oncologist

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Enzinger, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Moffitt Cancer Center, Tampa, Florida
  - Boston Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weeks JC, Catalano PJ, Cronin A, Finkelman MD, Mack JW, Keating NL, Schrag D. Patients' expectations about effects of chemotherapy for advanced cancer. N Engl J Med. 2012 Oct 25;367(17):1616-25. doi: 10.1056/NEJMoa1204410. PMID 23094723
- [Background] Degner LF, Sloan JA, Venkatesh P. The Control Preferences Scale. Can J Nurs Res. 1997 Fall;29(3):21-43. PMID 9505581
- [Background] Mazor KM, Street RL Jr, Sue VM, Williams AE, Rabin BA, Arora NK. Assessing patients' experiences with communication across the cancer care continuum. Patient Educ Couns. 2016 Aug;99(8):1343-8. doi: 10.1016/j.pec.2016.03.004. Epub 2016 Mar 6. PMID 26979476
- [Background] Legare F, Kearing S, Clay K, Gagnon S, D'Amours D, Rousseau M, O'Connor A. Are you SURE?: Assessing patient decisional conflict with a 4-item screening test. Can Fam Physician. 2010 Aug;56(8):e308-14. PMID 20705870
- [Background] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At the time of study closure, 5 participants were enrolled to usual care, 5 to the intervention arm.
Period: Overall Study
Arm/Group | Chemotherapy Education Intervention Arm | Usual Chemotherapy Education Arm
Started | 5 | 5
Completed (Early closure for failure to accrue) | 2 | 5
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy Education Intervention Arm | Usual Chemotherapy Education Arm | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Accurate Understanding of Chemotherapy Benefits at 8-12 Weeks
Description: Participants were asked how likely they thought chemotherapy was to cure their cancer (response options: very likely, somewhat likely, a little likely, not at all likely, don't know). Not at all likely is considered accurate, all other responses are considered inaccurate.
Time Frame: 8-12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Education Intervention Arm | Usual Chemotherapy Education Arm
Number analyzed (Participants) | 2 | 5
Participants | 0 | 0

2. Secondary Outcome: Understanding of Chemotherapy Risks
Description: Participants will be asked to rate the likelihood that they would experience specific side effects as a result of the chemotherapy under consideration (fatigue, nausea/vomiting, neuropathy, myalgias/arthralgias, hair loss, diarrhea). Patients' responses will be correlated to the known side effect profile of their chemotherapy regimen. Participants who are accurate on all questions will be considered to have accurate knowledge.
Time Frame: 2 weeks
Population: participants who completed the 2-week survey
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Education Intervention Arm | Usual Chemotherapy Education Arm
Number analyzed (Participants) | 3 | 5
Participants | 0 | 3

3. Secondary Outcome: Communication Satisfaction as Measured by 5 Items From the CAHPS Cancer Care Survey
Description: Communication satisfaction: will be assessed by five communication satisfaction items from the cancer specific version of the Consumer Assessment for Health Providers and Systems (CAHPS): "How often did your doctors...listen carefully to you, explain things in a way you could understand, give you as much information as you wanted about your cancer treatments, encourage you to ask all the questions you had, and treat you with courtesy and respect?" Options: always, usually, sometimes, or never. Patient responses will be summed, with possible score of 0-100 (with higher scores indicating better communication). Patients will complete this assessment at the post-decision and 3-month survey, but our primary analysis for this outcome will consider the post-decision assessment because it is most proximate to chemotherapy decision-making and exposure to the intervention.
Time Frame: 2 weeks
Population: Results are reported among the 5 patients in the usual care arm and 3 patients in the intervention arm that responded to this item on the 2-week survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chemotherapy Education Intervention Arm | Usual Chemotherapy Education Arm
Number analyzed (Participants) | 3 | 5
score on a scale | 90 (17.3) | 99 (2.24)

4. Secondary Outcome: Satisfaction With Chemotherapy Educational Materials Assessed on a 5-point Likert Scale.
Description: At the post-decision assessment, patients in the intervention arm will be asked to rate their satisfaction with the investigational chemotherapy educational materials with the following item: "Please think about the booklet, video, and website together. How would you rate them as a whole?" with response options on a 5-point likert scale where higher scores indicate greater satisfaction. (range: 1-5, 5 is best) Patients could alternatively choose "don't know, or I did not review them."
  Patients in the control arm will be asked to rate chemotherapy educational materials they were given with the same response options.
Time Frame: 2 weeks
Population: Analysis population includes participants who responded to this item on the 2-week survey. Of note, only 1 out of the 5 usual care participants responded to this question (presumably because they did not recall receiving any educational materials). 3 out of the 3 2-week survey respondents on the intervention arm responded to this item. The 3 reported satisfaction scores in the intervention arm were identical, hence a standard deviation of 0
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chemotherapy Education Intervention Arm | Usual Chemotherapy Education Arm
Number analyzed (Participants) | 3 | 1
score on a scale | 4 (0) | 3 (0)

5. Secondary Outcome: Decisional Conflict as Measured by the 4-item SURE
Description: Decisional conflict will be assessed by the SURE test of Legare et al, which includes 4 items assessing whether patients feel (yes/no) 1) sure of their decision, 2) understand benefits and risks of each option, 3) are clear about which risks and benefits matter most to them, and 4) if they have enough support for the decision. Scores range from 0-4, with lower scores indicating more decisional conflict. Scores of 3 or less are considered positive for the presence of decisional conflict.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chemotherapy Education Intervention Arm | Usual Chemotherapy Education Arm
Number analyzed (Participants) | 3 | 5
score on a scale | 3.67 (.58) | 3.8 (.45)

6. Secondary Outcome: Achievement of Preferred Role in Treatment Decision Making Process, as Measured by Degner's Control Preferences Scale
Description: Whether patients achieved their preferred role in decision-making will be assessed by the two-item Degner's Control Preferences Scale (CPS) which assesses and compares patients' preferred role (baseline) and achieved role (post-decision) decision-making.
  At baseline patients are asked so select among 5 options their preferred decision-making role - with two options representing an active role, two representing a passive role, and one representing shared decision-making. At post-decision, patients indicate what role they played in their treatment decision, with 5 similarly worded options representing active, passive, or shared decision-making.
  Patients whose preferred decision-making role (passive, shared, or active) matches their achieved role (passive, shared, or active) will be considered to have achieved their preferred role in their treatment decision.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Education Intervention Arm | Usual Chemotherapy Education Arm
Number analyzed (Participants) | 3 | 5
Participants | 2 | 3

7. Secondary Outcome: Decisional Regret
Description: Patient decisional regret will be assessed with Brehaut's 5-item Decisional Regret Scale. In this scale patients respond to a series of 5 questions about their recent treatment decision, with response options ranging from 1 (strongly agree) to 5 (strongly agree) on a 5-point likert scale. Two items are reverse-code, averaged, and converted to a 0-100 scale by subtracting 1 and multiplying by 25. A score of 100 indicates maximal regret.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Chemotherapy Education Intervention Arm | Usual Chemotherapy Education Arm
Number analyzed (Participants) | 2 | 5
score on a scale | 15 (7) | 7 (11)

8. Secondary Outcome: Discussions About End-of-life Care Preferences With Healthcare Proxy and Care Team
Description: At 8-12 weeks and 6 months, patients will indicate whether they have designated a healthcare proxy, or discussed end-of-life wishes with their physicians or proxy.
Time Frame: 3 months
Population: of the 2 patients in the intervention arm who completed the 3-month survey, neither had appointed a healthcare proxy; therefore, this question was skipped
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy Education Intervention Arm | Usual Chemotherapy Education Arm
Number analyzed (Participants) | 0 | 5
Participants | 0 | 5

ADVERSE EVENTS:
Time Frame: 6 months
Description: no SAEs occurred
Arm/Group | Chemotherapy Education Intervention Arm | Usual Chemotherapy Education Arm
All-Cause Mortality (participants affected / at risk) | 1/5 | 3/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
Study closed early for slow accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT03602885/Prot_SAP_000.pdf